CLINICAL TRIAL: NCT00309608
Title: A Randomised, Double-blind, Placebo-controlled, Five Parallel Groups Study Investigating the Efficacy and Safety of BI 1356 BS (1 mg, 5 mg and 10 mg Administered Orally Once Daily) Over 12 Weeks as add-on Therapy in Patients With Type 2 Diabetes and Insufficient Glycaemic Control Despite Metformin Therapy, Including an Open-label Glimepiride Treatment Arm.
Brief Title: Efficacy and Safety of BI 1356 BS (Linagliptin) in Combination With Metformin in Patients With type2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.6; 2005-004597-24 (EudraCT Number: EudraCT)
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Results first posted 2011-06-15 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; glimepiride

ARMS (5):
- Linagliptin low dose (Experimental): Patients receive Linagliptin low dose tablets once daily
  Interventions: Drug: Linagliptin
- Linagliptin medium dose (Experimental): Patients receive Linagliptin medium dose tablets once daily
  Interventions: Drug: Linagliptin
- Linagliptin high dose (Experimental): Patients receive Linagliptin high dose tablets once daily
  Interventions: Drug: Linagliptin
- Placebo (Placebo Comparator): Patients receive tablets identical to those containing Linagliptin low, medium and high dose
  Interventions: Drug: Placebo
- Glimepiride (Active Comparator): Patients receive Glimepiride tablets once daily
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Linagliptin — Linagliptin medium dose tablet once daily
  Arms: Linagliptin medium dose
Drug: Linagliptin — Linagliptin high dose tablet once daily
  Arms: Linagliptin high dose
Drug: Linagliptin — Linagliptin low dose tablet once daily
  Arms: Linagliptin low dose
Drug: Placebo — Placebo tablets once daily
  Arms: Placebo
Drug: Glimepiride — Glimepiride tablets once daily
  Arms: Glimepiride

SUMMARY:
The objective of the study is to test the efficacy, safety and tolerability of several doses of BI 1356 BS (1, 5, or 10 mg taken once daily) compared to placebo given for 12 weeks together with metformin in patients with type 2 diabetes mellitus who are not at goal with their HbA1c levels. In addition, there will be an unblinded treatment arm with glimepiride as add-on therapy to metformin for comparison. The influence of several factors (gender, age, weight, race, etc.) on the bioavailability and efficacy of BI 1356 BS will also be tested in this study.

ELIGIBILITY:
Inclusion criteria:

Inclusion_Criteria:

* Male and female patients with a diagnosis of type 2 diabetes mellitus and previo usly treated with metformin alone or with metformin and one other oral antidiabetic d rug
* HbA1c 7.0 9.0% at screening for patients treated with metformin and one other oral antidiabetic drug
* HbA1c 7.5 10.0% at screening for patients treated with metformin alone
* HbA1c 7.5 10.0% at beginning of the placebo run-in phase
* Age > 21 and < 75 years
* MI > 25 and < 40 kg/m2 (Body Mass Index)

Exclusion criteria:

Exclusion_Criteria:

* Clinically relevant cardiovascular disease
* Impaired hepatic function
* Renal insufficiency or impaired renal function
* Treatment with rosiglitazone or pioglitazone within 6 months prior to screening
* Treatment with insulin within 3 months prior to screening

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2006-04; Primary Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (48):
- France (5):
  - 1218.6.3302A Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.6.3303A Boehringer Ingelheim Investigational Site, Joué Les Tours
  - 1218.6.3304A Boehringer Ingelheim Investigational Site, Joué-lès-Tours
  - 1218.6.3305A Euraxi Pharma, Joué-lès-Tours
  - 1218.6.3301A Boehringer Ingelheim Investigational Site, Paris
- Germany (15):
  - 1218.6.49007 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 1218.6.49013 Boehringer Ingelheim Investigational Site, Bosenheim
  - 1218.6.49008 Boehringer Ingelheim Investigational Site, Dresden
  - 1218.6.49009 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1218.6.49014 Boehringer Ingelheim Investigational Site, Heidelberg
  - 1218.6.49012 Boehringer Ingelheim Investigational Site, Immenstadt im Allgäu
  - 1218.6.49001 Boehringer Ingelheim Investigational Site, Mainz
  - 1218.6.49005 Boehringer Ingelheim Investigational Site, Neuwied
  - 1218.6.49017 Boehringer Ingelheim Investigational Site, Offenbach A. M.
  - 1218.6.49002 Boehringer Ingelheim Investigational Site, Saarbrücken
  - 1218.6.49010 Boehringer Ingelheim Investigational Site, Saint Ingbert/Oberwürzbach
  - 1218.6.49011 Boehringer Ingelheim Investigational Site, Sinsheim
  - 1218.6.49015 Boehringer Ingelheim Investigational Site, Sulzbach-Rosenberg
  - 1218.6.49016 Boehringer Ingelheim Investigational Site, Wangen
  - 1218.6.49003 Boehringer Ingelheim Investigational Site, Würzburg
- Slovakia (4):
  - 1218.6.42103 Boehringer Ingelheim Investigational Site, Banská Bystrica
  - 1218.6.42104 Boehringer Ingelheim Investigational Site, Bratislava
  - 1218.6.42105 Boehringer Ingelheim Investigational Site, Bratislava
  - 1218.6.42101 Boehringer Ingelheim Investigational Site, Nové Mesto nad Váhom
- Sweden (4):
  - 1218.6.46003 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1218.6.46001 Boehringer Ingelheim Investigational Site, Malmo
  - 1218.6.46002 Boehringer Ingelheim Investigational Site, Uddevalla
  - 1218.6.46004 Boehringer Ingelheim Investigational Site, Uppsala
- Ukraine (4):
  - 1218.6.38002 Boehringer Ingelheim Investigational Site, Dnyepropetrovsk
  - 1218.6.38001 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.6.38003 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.6.38005 Boehringer Ingelheim Investigational Site, Kiev
- United Kingdom (16):
  - 1218.6.44012 Boehringer Ingelheim Investigational Site, Ashford
  - 1218.6.44004 Boehringer Ingelheim Investigational Site, Baillieston, Glasgow
  - 1218.6.44002 Boehringer Ingelheim Investigational Site, Bath
  - 1218.6.44003 Boehringer Ingelheim Investigational Site, Birmingham
  - 1218.6.44013 Boehringer Ingelheim Investigational Site, Camberley
  - 1218.6.44016 Boehringer Ingelheim Investigational Site, Chorley
  - 1218.6.44007 Boehringer Ingelheim Investigational Site, Dundee
  - 1218.6.44006 Boehringer Ingelheim Investigational Site, Exeter
  - 1218.6.44005 Boehringer Ingelheim Investigational Site, Gillingham
  - 1218.6.44015 Boehringer Ingelheim Investigational Site, Glasgow
  - 1218.6.44008 Boehringer Ingelheim Investigational Site, Guildford
  - 1218.6.44017 Boehringer Ingelheim Investigational Site, Liverpool
  - 1218.6.44001 Boehringer Ingelheim Investigational Site, London
  - 1218.6.44018 Boehringer Ingelheim Investigational Site, Manchester
  - 1218.6.44009 Boehringer Ingelheim Investigational Site, Newcastle upon Tyne
  - 1218.6.44019 Boehringer Ingelheim Investigational Site, Reading

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients randomized to receive treatment with matching placebo
- Linagliptin 1 mg: Patients randomized to receive treatment with Linagliptin 1 mg
- Linagliptin 5 mg: Patients randomized to receive treatment with Linagliptin 5 mg
- Linagliptin 10 mg: Patients randomized to receive treatment with Linagliptin 10 mg
- Glimepiride: Patients randomized to receive treatment with Glimepiride
Period: Overall Study
Arm/Group | Placebo | Linagliptin 1 mg | Linagliptin 5 mg | Linagliptin 10 mg | Glimepiride
Started | 71 | 65 | 66 | 66 | 65
Completed | 57 | 52 | 56 | 60 | 61
Not Completed | 14 | 13 | 10 | 6 | 4
Not completed — Adverse Event | 1 | 5 | 3 | 2 | 3
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 4 | 2 | 0 | 0
Not completed — Other incl. Lack of efficacy | 10 | 4 | 3 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linagliptin 1 mg | Linagliptin 5 mg | Linagliptin 10 mg | Glimepiride | Total
Number analyzed (Participants) | 71 | 65 | 66 | 66 | 65 | 333
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (8.1) | 59.2 (8.4) | 59.6 (9.8) | 61.8 (8.8) | 59.4 (9.9) | 60.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 29 | 31 | 24 | 140
  Male | 44 | 36 | 37 | 35 | 41 | 193
Body Mass Index (BMI) continuous [Mean (Standard Deviation); unit: kg/m^2] | 32.2 (4.2) | 32.3 (4.3) | 31.7 (4.5) | 31.7 (4.5) | 31.5 (4.2) | 31.9 (4.3)
Glycosylated Hemoglobin A1 (HbA1C) continuous [Mean (Standard Deviation); unit: Percent] | 8.37 (0.74) | 8.24 (0.74) | 8.46 (0.85) | 8.35 (0.73) | 8.22 (0.70) | 8.33 (0.75)
Fasting plasma glucose (FPG) continuous [Mean (Standard Deviation); unit: mg/dL] | 185.5 (38.8) | 182.3 (42.0) | 189.3 (42.4) | 188.7 (42.4) | 179.9 (40.4) | 185.1 (41.0)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline at Week 12
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 12 HbA1c percent minus the HbA1c percent baseline value. Means are treatment adjusted for baseline HbA1c.
Time Frame: Baseline and week 12
Population: The Full Analysis Set (FAS) included all treated and randomised patients with a baseline and at least one on-treatment HbA1c measurement available. Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin 1 mg | Linagliptin 5 mg | Linagliptin 10 mg | Glimepiride
Number analyzed (Participants) | 70 | 64 | 62 | 66 | 64
Percent | 0.25 (0.10) | -0.15 (0.10) | -0.48 (0.11) | -0.42 (0.10) | -0.59 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 10 mg; Linagliptin 10 mg vs. Placebo Missing endpoints after 12 weeks of treatment were replaced using "Last Observation Carried Forward" (LOCF); Test type: Superiority or Other; p < 0.0001, Pairwise comparison based on ANCOVA — There was no adjustment for multiple testing, however a hierarchy approach to control for the Type-I error was used. If the 10mg was not successful, any analysis of the 5mg will be descriptive, and similarly for the next step for the 1mg; Mean Difference (Final Values) = -0.67, 95% CI [-0.95 to -0.39], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo vs Linagliptin 5 mg; Linagliptin 5 mg vs. Placebo missing endpoints after 12 weeks of treatment were replaced using "Last Observation Carried Forward" (LOCF); Test type: Superiority or Other; p < 0.0001, Pairwise comparison based on ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.73, 95% CI [-1.01 to -0.44], Standard Error of Mean 0.14
Statistical Analysis 3: Comparison: Placebo vs Linagliptin 1 mg; Linagliptin 1 mg vs. Placebo Missing endpoints after 12 weeks of treatment were replaced using "Last Observation Carried Forward" (LOCF); Test type: Superiority or Other; p = 0.0055, Pairwise comparison based on ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI [-0.68 to -0.12], Standard Error of Mean 0.14
Statistical Analysis 4: Comparison: Placebo vs Linagliptin 10 mg; Placebo vs. Linagliptin 10 mg Analysis additionally adjusted for previous anti-diabetic medication. Missing endpoints after 12 weeks of treatment were replaced using Last Observation Carried Forward (LOCF); Test type: Superiority or Other; p < 0.0001, Pairwise comparison based on ANCOVA; Mean Difference (Final Values) = -0.73, 95% CI [-0.99 to -0.46], Standard Error of Mean 0.14
Statistical Analysis 5: Comparison: Placebo vs Linagliptin 5 mg; Linagliptin 5 mg vs. Placebo Analysis additionally adjusted for previous anti-diabetic medication. Missing endpoints after 12 weeks of treatment were replaced using "last observation carried forward" (LOCF); Test type: Superiority or Other; p < 0.0001, Pairwise comparison based on ANCOVA; Mean Difference (Final Values) = -0.75, 95% CI [-1.02 to -0.48], Standard Error of Mean 0.14
Statistical Analysis 6: Comparison: Placebo vs Linagliptin 1 mg; Linagliptin 1 mg vs. Placebo Analysis additionally adjusted for previous anti-diabetic medication. Missing endpoints after 12 weeks of treatment were replaced using "last observation carried forward" (LOCF); Test type: Superiority or Other; p = 0.0049, Pairwise comparison based on ANCOVA; Mean Difference (Final Values) = -0.39, 95% CI [-0.66 to -0.12], Standard Error of Mean 0.14

2. Secondary Outcome: Percentage of Patients With HbA1c<=7.0% at Week 12
Description: Descriptive calculation of Patients with HbA1c <= 7.0% at Week 12.
Time Frame: week 12
Population: This population includes the Full Analysis Set (FAS). Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Number; unit: Percentage of Patients
Arm/Group | Placebo | Linagliptin 1 mg | Linagliptin 5 mg | Linagliptin 10 mg | Glimepiride
Number analyzed (Participants) | 70 | 64 | 62 | 66 | 64
Percentage of Patients | 1.4 | 15.6 | 14.5 | 21.2 | 31.3
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 10 mg; Linagliptin 10 mg vs. Placebo; Test type: Superiority or Other; p = 0.0054, Regression, Logistic; Odds Ratio (OR) = 18.575, 95% CI 2-sided [2.367 to 145.781]
Statistical Analysis 2: Comparison: Placebo vs Linagliptin 5 mg; Linagliptin 5 mg vs. Placebo; Test type: Superiority or Other; p = 0.0214, Regression, Logistic; Odds Ratio (OR) = 11.715, 95% CI 2-sided [1.439 to 95.351]
Statistical Analysis 3: Comparison: Placebo vs Linagliptin 1 mg; Linagliptin 1 mg vs. Placebo; Test type: Superiority or Other; p = 0.0167, Regression, Logistic; Odds Ratio (OR) = 12.776, 95% CI 2-sided [1.586 to 102.895]
Statistical Analysis 4: Comparison: Placebo vs Glimepiride; Glimepiride vs. Placebo; Test type: Superiority or Other; p = 0.0010, Regression, Logistic; Odds Ratio (OR) = 31.360, 95% CI 2-sided [4.063 to 242.028]

3. Secondary Outcome: Fasting Blood Plasma Glucose Level (FPG) Change From Baseline at Week 12
Description: This change from baseline reflects the Week 12 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 12
Population: This population includes the FAS using the LOCF imputation, with the further restriction of patients with a baseline and post-baseline FPG value.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin 1 mg | Linagliptin 5 mg | Linagliptin 10 mg
Number analyzed (Participants) | 68 | 63 | 62 | 66
mg/dL | 13.63 (4.30) | -5.32 (4.51) | -21.29 (4.48) | -15.87 (4.33)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 10 mg; Linagliptin 10mg vs. Placebo; Test type: Superiority or Other; p < 0.0001, Pairwise comparison based on ANCOVA; Mean Difference (Final Values) = -29.5, 95% CI [-41.4 to -17.5], Standard Error of Mean 6.07
Statistical Analysis 2: Comparison: Placebo vs Linagliptin 5 mg; Linagliptin 5mg vs. Placebo; Test type: Superiority or Other; p < 0.0001, Pairwise comparison based on ANCOVA; Mean Difference (Final Values) = -34.92, 95% CI [-47.0 to -22.8], Standard Error of Mean 6.16
Statistical Analysis 3: Comparison: Placebo vs Linagliptin 1 mg; Linagliptin 1 mg vs. Placebo; Test type: Superiority or Other; p = 0.0022, Pairwise comparison based on ANCOVA; Mean Difference (Final Values) = -18.95, 95% CI [-31.0 to -6.87], Standard Error of Mean 6.13

ADVERSE EVENTS:
Time Frame: 12 Weeks + 30 Days
Description: MedDRA version 10.0 was used for reporting.
Arm/Group | Placebo | Linagliptin 1 mg | Linagliptin 5 mg | Linagliptin 10 mg | Glimepiride
Serious Adverse Events (participants affected / at risk) | 1/71 | 3/65 | 1/66 | 4/66 | 1/65
Other Adverse Events (participants affected / at risk) | 10/71 | 4/65 | 8/66 | 8/66 | 4/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=71) | Linagliptin 1 mg (N=65) | Linagliptin 5 mg (N=66) | Linagliptin 10 mg (N=66) | Glimepiride (N=65)
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal mass (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=71) | Linagliptin 1 mg (N=65) | Linagliptin 5 mg (N=66) | Linagliptin 10 mg (N=66) | Glimepiride (N=65)
Nausea (Gastrointestinal disorders) | 3 | 0 | 4 | 3 | 0
Nasopharyngitis (Infections and infestations) | 7 | 4 | 5 | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.